CLINICAL TRIAL: NCT05906849
Title: Where We All Meet: ACT as a Conceptual and Therapeutic Transdiagnostic Approach to Adolescents With Different Anxiety Disorders
Brief Title: Where We All Meet: ACT Approach to Adolescents Anxiety Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Diana Vieira Figueiredo, M.Sc., University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.13986.BD
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Social Anxiety Disorder; Generalized Anxiety Disorder
Keywords: Acceptance and Commitment Therapy; Transdiagnostic Processes; Psychological Flexibility/Inflexibility; Adolescents; Anxiety Disorders
MeSH Terms: conditions — Phobia, Social; Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: To attain this project's aims a longitudinal research will take place. Adolescents presenting SAD or GAD will be randomly allocated to a Control Group (no intervention group), or an Experimental Group (individual intervention group). Adolescents with SAD will be randomly allocated to the control group (n≥13), and to the SAD Experimental Group (n=29). Similarly, adolescents with GAD will be randomly allocated to the control group (n≥13), the to the GAD Experimental Group (n=29). Therefore, the Randomized and Parallel Controlled Trial will include a Control Group (N=29), a SAD (n=29) and a GAD (n=29) Experimental Group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Group of participants with a main diagnosis of social anxiety disorder (n≥13) or generalized anxiety disorder (n≥13) not subjected to any psychological intervention within the current trial. They will be asked to fill in the self-report protocol at 2 different time points (12 weeks interval) mimicking the pre- and post-intervention assessment moments; these adolescents will be assessed after the second time point and referred to the school psychology services if the difficulties persist.
- SAD Intervention Group (Experimental): Group of participants with a main diagnosis of social anxiety disorder (n=26) subjected to individual online delivered 12 sessions ACT psychotherapy. Participants pertaining to this group will be assessed at 4 different time points (pre- and post-treatment and at a 3- and 6- month follow-up).
  Interventions: Behavioral: ACT for anxiety disorders
- GAD Intervention Group (Experimental): Group of participants with a main diagnosis of generalized anxiety disorder (n=26) subjected to individual online delivered 12 sessions ACT psychotherapy. Participants pertaining to this group will be assessed at 4 different time points (pre- and post-treatment and at a 3- and 6- month follow-up).
  Interventions: Behavioral: ACT for anxiety disorders

INTERVENTIONS:
Behavioral: ACT for anxiety disorders — A twelve session Acceptance and Commitment Therapy (ACT) for anxiety disorders, applied individually and remotely (through videoconference) to participants fulfilling inclusion criteria (i.e., participants included in the SAD and GAD Experimental Groups).
  Arms: GAD Intervention Group; SAD Intervention Group

SUMMARY:
Transdiagnostic approaches have been proposed as more truthfully representing mental health problems. Acceptance and Commitment Therapy (ACT) is a transdiagnostic approach that proposes Psychological Inflexibility/Flexibility (PI/PF) as the root of human suffering/flourishing. ACT has been recognized as conceptually and clinically relevant for adult disorders. However, during adolescence, when anxiety disorders are highly prevalent, the same evidence is scarce. Specifically, methodologically robust designs investigating ACT's efficacy on adolescents' ADs are scarce and mechanisms underlying change during ACT for adolescents with ADs have not been investigated. Therefore, this study aims to adapt, implement, and investigate the efficacy of an online delivered (through videoconference) ACT intervention to adolescents presenting SAD or GAD, thus contributing to amplifying the transdiagnostic application of ACT to these disorders. A Randomized Controlled Trial (RCT) with 3 groups (i.e., Control, GAD intervention, and SAD intervention groups) of adolescents aged between 14 and 18 years old will be conducted. Outcome measurement will be assessed at pre-intervention, post-intervention, and at 3- and 6-month follow-ups. The investigators expect improvements in outcome variables (e.g., anxiety symptoms) at post-treatment for intervention groups. When comparing changes in outcome variables between the control and the intervention groups, improvements are expected only in the groups receiving intervention. Additionally, similar effects on outcome measures are expected in both intervention groups with gains being maintained over time (i.e., at 3- and 6-months follow-up). Finally, changes in PI/PF processes are expected to predict changes in outcome variables in both intervention groups. This RCT will provide valuable insights that can potentially enhance the efficacy of treatment modalities, contributing to improved well-being for adolescents with ADs.

DETAILED DESCRIPTION:
Recently, researchers have increasingly focused on understanding commonalities in psychological processes underlying human suffering and psychopathology [1,2]. This has been driven by multiple factors, namely: high comorbidity among mental health problems [e.g., 3,4]; evidence for within-disorder and between-disorder prediction and cascading effects throughout life [e.g., 5,6]; data suggesting that disorder-specific interventions produce improvements in comorbid disorders [e.g., 7,8]; established efficacy of transdiagnostic interventions in multiple disorders [e.g., 9,10]; and their equivalent efficacy to diagnosis-specific interventions [11]. Taken together, research indicates the presence of shared mechanisms, highlighting the need for treatments to target broader processes. Accordingly, transdiagnostic approaches have emerged as promising frameworks, as they may better reflect the complexity and dimensionality of the human experience and more accurately represent the reality of mental health problems.

Acceptance and Commitment Therapy (ACT) is a transdiagnostic approach to behavior change that proposes Psychological Inflexibility (PI) as the root of human suffering in general, and of mental health disorders in particular [12]. PI is defined as rigid attempts to control, alter or minimize unpleasant internal experiences at the expense of the ability to persist and/or change behavior to pursue chosen values. PI steams from six interrelated processes: Cognitive Fusion, Experiential Avoidance, Attachment to the Conceptualized Self, Dominance of the Conceptualized Past/Feared Future, Lack of Values Clarity and Inaction, Impulsivity or Avoidant Persistence [13]. ACT aims to reverse PI processes by cultivating Psychological Flexibility (PF) which refers to the ability to be in contact with the present moment regardless of unpleasant internal experiences while persisting in value-guided behaviors [14]. PF entails six interrelated processes, opposing each PI processes: Cognitive Defusion, Acceptance, Self as Context, Contact with the Present Moment, Values, and Committed Action [12].

Evidence supports ACT's efficacy in adults with various disorders [e.g.,15, 16] as well as the role of PI/PF components as mechanisms of change following ACT [17]. Some studies support that role in adolescents' mental health [18,19] and promising results suggest ACT's efficacy with this population [e.g.,20]. However, most studies did not consider all PI/PF processes [e.g., 21] and there is a scarcity of methodologically robust designs (e.g., Randomized Controlled Trials; RCTs) investigating ACT interventions in adolescents [e.g.,10]. Because most studies did not include extended follow-ups and adolescence is marked by significant and rapid psychological changes [22], ACT's utility to this age group has not been fully assessed. This seems worrisome considering that between 10 to 20% of adolescents experience mental health problems [23]. In youth, anxiety disorders are the most common disorders [24]. Particularly, Social Anxiety Disorder (SAD) and Generalized Anxiety Disorder (GAD) present significant prevalence rates in adolescents [4,25] both typically presenting a chronic course that may evolve into other mental health disorders in adulthood [6,26]. ACT has been proven effective for SAD and GAD treatment in adults [27,28]. Preliminary findings point to ACT being efficacious for treating anxiety in adolescence [23]. However, few studies examined ACT's efficacy for adolescents' SAD [20,29], and only one included adolescents with GAD [20]. Research on the efficacy of ACT to adolescents' SAD and GAD is largely missing, and mechanisms underlying change have not been reported. Increasing the understanding of the common mechanisms underlying mental health problems in adolescents, and how these mechanisms can be used to sustain efficacious psychological interventions, is a crucial research concern.

Thus, this project intends to amplify the transdiagnostic application of ACT to adolescents presenting SAD and GAD. A RCT will be conducted to explore the efficacy and processes of change of ACT for SAD or GAD, considering adolescents' anxiety symptoms and flourishing as outcomes. The research team will adapt, implement, and investigate the efficacy of an online delivered (videoconference) ACT Intervention to adolescents presenting SAD or GAD via: : 1. Changes in primary (i.e., anxiety symptoms) and secondary (i.e., flourishing and PI/PF processes) outcomes following intervention - significant improvements are expected at post-intervention only in the intervention groups (i.e., SAD intervention and GAD intervention groups), in comparison with a clinical control group; 2. Examining the stability of change over time (i.e., 3- and 6-months follow-up) - improvements are expected to maintain; 3. Comparing the efficacy of the intervention between both intervention groups - Similar effects on outcome measures for both clinical groups are expected; 4. Investigating mechanisms of change following intervention in both intervention groups - Similar findings in both intervention groups are expected, with changes in PI/PF predicting changes in outcome variables.

All procedures involved in this project (described elsewhere in this form) were approved by the Ethics Committee of the Faculty of Psychology and Educational Sciences, University of Coimbra and the General Directorate of Education authorized the data collection protocol to be implemented in school contexts. Informed consent from adolescents and their parents/legal guardians will be required for all potential participants prior to any data collection. Adolescents and their parents/legal guardians will be informed that the participation is voluntary and that they can decline to participate at any time during the project without any negative consequence. Moreover, they will be informed that the confidentiality of responses will be assured in all moments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescent's sample: No mental health diagnosis;
* Adolescents with SAD sample: Main diagnosis of SAD;
* Adolescents with GAD sample: Main diagnosis of GAD. Note: adolescents presenting both GAD and SAD will be excluded as its inclusion could confound the projects' results and conclusions.

Exclusion criteria:

1. Cognitive impairment (assessed through a clinical interview; MINI-KID [37,38]);
2. Presence of psychotic symptoms or suicidal ideation (according to the MINI-KID [37,38]);
3. Undergoing another treatment (e.g., medication) for a psychiatric condition.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Social Anxiety and Avoidance Scale for Adolescents | Baseline, Week 12, Follow-Up 3 Months and Follow-Up 6 Months
  The SAASA consists of 30 items in its adapted version for late adolescents [30]. It intends to assess the degree of anxiety and frequency of avoidance in social situations representative of the most frequent social fears during adolescence. Each item (e.g., "Going to a party given by a colleague") is answered twice, for two subscales - anxiety and avoidance -, on a five-point Likert scale (ranging from 1 = 'none' to 5 = 'very much' for anxiety; and from 1 = 'never' to 5 = 'almost always' for avoidance). Previous psychometric information indicates very good internal consistency values, convergent validity in relation to other measures of anxious and depressive symptoms, and measurement invariance across gender and age [30, 31]
Change in Generalized Anxiety Disorder - 7 | Baseline, Week 12, Follow-Up 3 Months and Follow-Up 6 Months
  The GAD-7 [32,33] is a 7 item self-report scale initially designed to identify probable cases of Generalized Anxiety Disorder (GAD). The GAD-7 assesses Generalized Anxiety Disorder symptoms such as nervousness, uncontrollability of worry, excessive worry, restlessness, difficulty in relaxing and easy irritability. Items (e.g., "Feeling nervous, anxious or on edge") are answered in 4-point Liker scale (ranging from 0='not at all' to 3= 'nearly every day') reporting to the two previous weeks. Higher scores on the GAD-7 represent higher levels of GAD symptoms. Previous psychometric information indicates excellent internal consistency values and divergent validity in relation to measures of quality of life and satisfaction with school [33].

SECONDARY OUTCOMES:
Change in the Multidimensional Psychological Flexibility Inventory - 24 (short form) | Baseline, Week 12, Follow-Up 3 Months and Follow-Up 6 Months
  The MPFI-24 [34] is a 24-item self-report scale for the assessment of psychological flexibility/inflexibility, comprised by 12 subscales, representing psychological flexibility (i.e., Acceptance, Present Moment Awareness, Self as Context, Defusion, Values, Committed Action) and psychological inflexibility (i.e., Experiential Avoidance, Lack of Contact with the Present Moment, Self as Content, Fusion, Lack of Contact with Values, Inaction). Items (e.g., "I opened myself to all of my feelings, the good and the bad") are answered on a 6-point Likert scale (ranging from 1 = 'never true' to 6 = 'always true') reporting to the previous 2 weeks. The scores of the 6 flexibility and 6 inflexibility subscales can be averaged to create a composite score representing global flexibility and inflexibility, respectively. Previous psychometric information indicates good to excellent internal consistency values [34] . This measure is currently being adapted and validated to Portuguese adolescents.
Change in Mental Health Continuum - Short Form - for youth | Baseline, Week 12, Follow-Up 3 Months and Follow-Up 6 Months
  The MHC-SF [35,36] is a 14 items self-report measure that assesses adolescent's flourishing based on levels of subjective well-being across 3 domains: emotional, social and psychological well-being. Following the instructions (i.e., "Please answer the following questions about how you have been feeling during the past month"), items (e.g., "How often do you felt happy?") are answered on a 6-points Likert scale (ranging from 0='Never' to 5='Every day'). Previous psychometric information indicates good internal consistency values and construct validity in relation to measures of quality of life, life satisfaction, anxiety, depression and internalizing and externalizing problems [36] .

CONTACTS AND LOCATIONS:
Overall Officials: Diana V Figueiredo, M.Sc., Principal Investigator — Center for Research in Neuropsychology and Cognitive and Behavioral Intervention (CINEICC), FPCE-UC
Locations (1):
- Center for Research in Neuropsychology and Cognitive and Behavioral Intervention (CINEICC), Faculty of Psychology and Educational Sciences - University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levin ME, MacLane C, Daflos S, Seeley J, Hayes SC, Biglan A, Pistorello J. Examining psychological inflexibility as a transdiagnostic process across psychological disorders. J Contextual Behav Sci. 2014 Jul;3(3):155-163. doi: 10.1016/j.jcbs.2014.06.003. PMID 29057212
- [Background] [2] Norton, P. (Ed.). (2017). Transdiagnostic Approaches [Special Issue]. 46. https://doi.org/10.1016/j.janxdis.2017.02.004
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Niermann HCM, Voss C, Pieper L, Venz J, Ollmann TM, Beesdo-Baum K. Anxiety disorders among adolescents and young adults: Prevalence and mental health care service utilization in a regional epidemiological study in Germany. J Anxiety Disord. 2021 Oct;83:102453. doi: 10.1016/j.janxdis.2021.102453. Epub 2021 Jul 10. PMID 34303082
- [Background] Asselmann E, Wittchen HU, Lieb R, Beesdo-Baum K. Sociodemographic, clinical, and functional long-term outcomes in adolescents and young adults with mental disorders. Acta Psychiatr Scand. 2018 Jan;137(1):6-17. doi: 10.1111/acps.12792. Epub 2017 Aug 31. PMID 28861892
- [Background] Copeland WE, Shanahan L, Costello EJ, Angold A. Childhood and adolescent psychiatric disorders as predictors of young adult disorders. Arch Gen Psychiatry. 2009 Jul;66(7):764-72. doi: 10.1001/archgenpsychiatry.2009.85. PMID 19581568
- [Background] Allen LB, White KS, Barlow DH, Shear MK, Gorman JM, Woods SW. Cognitive-Behavior Therapy (CBT) for Panic Disorder: Relationship of Anxiety and Depression Comorbidity with Treatment Outcome. J Psychopathol Behav Assess. 2010 Jun;32(2):185-192. doi: 10.1007/s10862-009-9151-3. Epub 2009 Jul 24. PMID 20421906
- [Background] [8] Tsao, J. C. I., Mystkowski, J. L., Zucker, B. G., & Craske, M. G. (2002). Effects of cognitive-behavioral therapy for panic disorder on comorbid conditions: Replication and extension. Behavior Therapy, 33(4), 493-509. https://doi.org/10.1016/S0005-7894(02)80013-2
- [Background] Powers MB, Zum Vorde Sive Vording MB, Emmelkamp PM. Acceptance and commitment therapy: a meta-analytic review. Psychother Psychosom. 2009;78(2):73-80. doi: 10.1159/000190790. Epub 2009 Jan 14. PMID 19142046
- [Background] [10] Petersen, J. M., Ona, P. Z., & Twohig, M. P. (2022). A Review of Acceptance and Commitment Therapy for Adolescents: Developmental and Contextual Considerations. Cognitive and Behavioral Practice. https://doi.org/10.1016/j.cbpra.2022.08.002
- [Background] Dalgleish T, Black M, Johnston D, Bevan A. Transdiagnostic approaches to mental health problems: Current status and future directions. J Consult Clin Psychol. 2020 Mar;88(3):179-195. doi: 10.1037/ccp0000482. PMID 32068421
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] [13] Hayes, S. C., Strosahl, K. D., & Wilson, K. G. (1999). Acceptance and commitment therapy: An experiential approach to behavior change (pp. xvi, 304). Guilford Press.
- [Background] [14] Hayes, S. C., Pistorello, J., & Levin, M. E. (2012). Acceptance and Commitment Therapy as a Unified Model of Behavior Change. The Counseling Psychologist, 40(7), 976-1002. https://doi.org/10.1177/0011000012460836
- [Background] [15] Gloster, A. T., Walder, N., Levin, M. E., Twohig, M. P., & Karekla, M. (2020). The empirical status of acceptance and commitment therapy: A review of meta-analyses. Journal of Contextual Behavioral Science, 18, 181-192.
- [Background] [16] García, L., & Valdivia-Salas, S. (2018). Efficacy of ACT on social anxiety disorder: A systematic review. Behavioral Psychology, 26, 247-260.
- [Background] Stockton D, Kellett S, Berrios R, Sirois F, Wilkinson N, Miles G. Identifying the Underlying Mechanisms of Change During Acceptance and Commitment Therapy (ACT): A Systematic Review of Contemporary Mediation Studies. Behav Cogn Psychother. 2019 May;47(3):332-362. doi: 10.1017/S1352465818000553. Epub 2018 Oct 4. PMID 30284528
- [Background] [18] Cobos-Sánchez, L., Flujas-Contreras, J. M., & Becerra, I. G. (2020). Relation between psychological flexibility, emotional intelligence and emotion regulation in adolescence. Current Psychology. https://doi.org/10.1007/s12144-020-01067-7
- [Background] Ciarrochi J, Kashdan TB, Leeson P, Heaven P, Jordan C. On being aware and accepting: a one-year longitudinal study into adolescent well-being. J Adolesc. 2011 Aug;34(4):695-703. doi: 10.1016/j.adolescence.2010.09.003. Epub 2010 Oct 14. PMID 20950848
- [Background] Hancock KM, Swain J, Hainsworth CJ, Dixon AL, Koo S, Munro K. Acceptance and Commitment Therapy versus Cognitive Behavior Therapy for Children With Anxiety: Outcomes of a Randomized Controlled Trial. J Clin Child Adolesc Psychol. 2018 Mar-Apr;47(2):296-311. doi: 10.1080/15374416.2015.1110822. Epub 2016 Mar 21. PMID 26998803
- [Background] [21] Lønfeldt, N. N., Silverman, W. K., & Esbjørn, B. H. (2017). A Systematic Review and Meta-analysis of the Association Between Third-Wave Cognitive Constructs and Youth Anxiety. Https://Doi.Org/10.1521/Ijct.2017.10.2.115. https://doi.org/10.1521/ijct.2017.10.2.115
- [Background] Christie D, Viner R. Adolescent development. BMJ. 2005 Feb 5;330(7486):301-4. doi: 10.1136/bmj.330.7486.301. No abstract available. PMID 15695279
- [Background] [23] World Health Organization. (2021, November 17). Adolescent mental health. https://www.who.int/news-room/fact-sheets/detail/adolescent-mental-health
- [Background] Merikangas KR, He JP, Burstein M, Swanson SA, Avenevoli S, Cui L, Benjet C, Georgiades K, Swendsen J. Lifetime prevalence of mental disorders in U.S. adolescents: results from the National Comorbidity Survey Replication--Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):980-9. doi: 10.1016/j.jaac.2010.05.017. Epub 2010 Jul 31. PMID 20855043
- [Background] Georgiades K, Duncan L, Wang L, Comeau J, Boyle MH; 2014 Ontario Child Health Study Team. Six-Month Prevalence of Mental Disorders and Service Contacts among Children and Youth in Ontario: Evidence from the 2014 Ontario Child Health Study. Can J Psychiatry. 2019 Apr;64(4):246-255. doi: 10.1177/0706743719830024. PMID 30978138
- [Background] Ferdinand RF, Dieleman G, Ormel J, Verhulst FC. Homotypic versus heterotypic continuity of anxiety symptoms in young adolescents: evidence for distinctions between DSM-IV subtypes. J Abnorm Child Psychol. 2007 Jun;35(3):325-33. doi: 10.1007/s10802-006-9093-0. Epub 2007 Jan 17. PMID 17226094
- [Background] [27] Avdagic, E., Morrissey, S. A., & Boschen, M. J. (2014). A Randomised Controlled Trial of Acceptance and Commitment Therapy and Cognitive-Behaviour Therapy for Generalised Anxiety Disorder. Behaviour Change, 31(2), 110-130.
- [Background] [28] García-Pérez, L., & Valdivia-Salas, S. (2018). Intervención en el trastorno de ansiedad social a través de la terapia de aceptación y compromiso: Una revisión sistemática. [Acceptance and commitment therapy for social anxiety disorder: A systematic review.]. Behavioral Psychology, 26(2), 379-392.
- [Background] Azadeh SM, Kazemi-Zahrani H, Besharat MA. Effectiveness of Acceptance and Commitment Therapy on Interpersonal Problems and Psychological Flexibility in Female High School Students With Social Anxiety Disorder. Glob J Health Sci. 2015 Jul 12;8(3):131-8. doi: 10.5539/gjhs.v8n3p131. PMID 26493425
- [Background] [30] Vagos, P., Pereira, A., & Cunha, M. (2013). Evaluating social fears in late adolescence: Study with a Portuguese sample. European Journal of Developmental Psychology, 11(3), 373-385. https://doi.org/10.1080/17405629.2013.841093
- [Background] [31] Cunha, M., Pinto-Gouveia, J. P., & Salvador, M. C. (2008). Social fears in adolescence - The social anxiety and avoidance scale for adolescents. European Psychologist, 13, 197-213. https://doi.org/10.1027/1016-9040.13.3.197
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] [33] Gonçalves, M. (2019). Ansiedade em Crianças e Adolescentes - Validação da Escala GAD-7. [Master Dissertation, University of Coimbra]. Estudo Geral Repositório científico da UC. http://hdl.handle.net/10316/89592
- [Background] Rolffs JL, Rogge RD, Wilson KG. Disentangling Components of Flexibility via the Hexaflex Model: Development and Validation of the Multidimensional Psychological Flexibility Inventory (MPFI). Assessment. 2018 Jun;25(4):458-482. doi: 10.1177/1073191116645905. Epub 2016 May 5. PMID 27152011
- [Background] [35] Keyes, C. L. M. (2009). The Nature and Importance of Positive Mental Health in America's Adolescents. In R. Gilman, E. S. Huebner, & M. J. Furlong (Eds.), Handbook of positive psychology in schools (pp. 9-23). Routledge.
- [Background] [36] Matos, A. P., André, R. S., Cherpe, S., Rodrigues, D., Figueira, C., & Pinto, A. M. (2010). Estudo Psicométrico preliminar da Mental Health Continuum - Short Form - for youth numa amostra de adolescentes portugueses. Psychologica, 53, 131-156. https://doi.org/10.14195/1647-8606_53_7
- [Background] Sheehan DV, Sheehan KH, Shytle RD, Janavs J, Bannon Y, Rogers JE, Milo KM, Stock SL, Wilkinson B. Reliability and validity of the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID). J Clin Psychiatry. 2010 Mar;71(3):313-26. doi: 10.4088/JCP.09m05305whi. PMID 20331933
- [Background] [38] Ribeiro da Silva, D., Vagos, P. Brazão, N., & Rijo, D. (2017). Mini-Kid - Portuguese version. Unpublished material.